CLINICAL TRIAL: NCT05787834
Title: Respiratory Muscle Training During Breast Cancer Treatment: Effects on the Autonomic Nervous System and Cardiotoxicity
Brief Title: Home-based Respiratory Muscle Training for Minimizing Side Effects in Patients Undergoing Treatment for Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I-3364822; NCI-2023-01256 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3364822 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2023-02-23; First posted 2023-03-28 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (low resistance RMT Group) (Active Comparator): Patients receive usual care for 12 weeks on study and a Respiratory Muscle training Device with small breathing resistance
  Interventions: Other: Best Practice; Other: Medical Device Usage and Evaluation; Procedure: Respiratory Muscle Training; Other: Survey Administration
- Group II (Moderate to highter resistance RMT) (Experimental): Patients undergo RMT using a respiratory muscle training device with moderate to higher breathing resistance for 12 weeks on study.
  Interventions: Other: Medical Device Usage and Evaluation; Procedure: Respiratory Muscle Training; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group I (low resistance RMT Group)
Other: Medical Device Usage and Evaluation — Wear accelerometer
Procedure: Respiratory Muscle Training — Undergo RMT
  Other Names: RMT
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates whether home-based respiratory muscle training is useful for minimizing side effects in patients undergoing treatment for breast cancer. Over-activation of the nervous system during breast cancer treatment can result in heart- and lung-related side effects which have the potential to reduce a patient's quality of life. Aerobic exercise can help prevent the development of these side effects. However, engaging in regular aerobic exercise may be difficult for breast cancer patients who are actively undergoing treatment. Respiratory muscle training (RMT) involves a series of breathing and other exercises that are performed to improve the function of the respiratory muscles through resistance and endurance training. Home-based RMT may represent a more feasible approach for reducing side effects in patients undergoing treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility of delivering a 12-week RMT program during adjuvant and neoadjuvant chemotherapy used to treat breast cancer.

SECONDARY OBJECTIVES:

I. To determine how cardiac autonomic regulation, cardiorespiratory fitness, exercise performance, and quality-of-life (QoL) are affected by RMT during breast cancer treatment.

II. To assess how RMT affects patient reported symptoms linked to sympathetic overactivation such as stress, fatigue, dyspnea, when performed during chemotherapy.

EXPLORATORY OBJECTIVE:

I. To determine if RMT reduces circulating biomarkers of autonomic dysfunction, inflammation, and cardiac injury in breast cancer patients undergoing treatment.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: patients receive lower resistance RMT using a respiratory muscle training device for 12 weeks.

GROUP II: Patients undergo higher resistance RMT using a respiratory muscle training device for 12 weeks on study.

ELIGIBILITY:
Inclusion Criteria:

* Documented breast cancer and scheduled to receive adjuvant or neoadjuvant chemotherapy
* Age >= 18 years old
* Cognitively capable of following direction and performing the intervention
* Able to speak, read and comprehend English language
* Understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, heart failure or psychiatric illness/social situations that would limit compliance with study requirements
* Prior radiation to the left chest wall
* Patients with medical frailty (clinical discretion)
* Are pregnant or nursing
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2028-10-16 (Estimated); Study Completion 2029-10-16 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who participate in the study | Up to 12 weeks
Proportion of patients who remain on study | Up to 12 weeks
Proportion of patients who perform >= 3 respiratory muscle training (RMT) sessions/week | Up to 12 weeks
  Overall compliance rates (compliance at all time points) will be estimated using 90% confidence intervals. Additionally, compliance status will be modeled as a function of time (e.g., week), and pre-specified exogenous factors (e.g., baseline age, performance status, self-reported history of exercise, breast cancer (BC) treatment received, treatment side-effects) using a generalized estimating equation (GEE) logistic regression model (auto-regressive covariance structure). Estimates of compliance rates will be obtained by time-point and tests about the appropriate contrasts of model estimates will be used to determine if there is a time trend.
Proportion of patients who perform > 70% of their RMT sessions | Up to 12 weeks
  Adherence rates (completion of >= 70% of sessions) will be estimated using 90% confidence intervals. Additionally, compliance status will be modeled as a function of time (e.g., week), and pre-specified exogenous factors (e.g., baseline age, performance status, self-reported history of exercise, BC treatment received, treatment side-effects) using a GEE logistic regression model (auto-regressive covariance structure). Estimates of compliance rates will be obtained by time-point and tests about the appropriate contrasts of model estimates will be used to determine if there is a time trend.

SECONDARY OUTCOMES:
Change in Functional Capacity | At baseline, 6 weeks, and 12 weeks
  Six minute walking test is a functional test of sub-maximum cardiorespiratory capacity.
Change in Lower body strength | At baseline, 6 weeks, and 12 weeks
  The Short Physical Performance Battery - PPB is comprised of 3 tasks: a hierarchial standing balance test (side by side, semi-tandem and tandem), 4-m habitual gait speed, and 5 sit to stand from a chair. Each task is scored (based on time) from 0-4 Points (p) and then summarized into a total score of 0-12 p, where 12 p represents the highest performance.
Assess Dyspnea | At baseline, 6 weeks, and 12 weeks
  Dyspnea will be measured by the Dyspnea-12 questionnaire which contains 12 items on a scale of 0(none), mild (1) and Severe (3) and evaluates the physical and affective dimensions of dyspnea. Higher scores represent greater severity.
Assess Fatigue | At baseline, 6 weeks, and 12 weeks
  Fatigue will be measured using the Brief Fatigue Inventory (BFI). Each item is scored 1 (no fatigue) to 10 (as bad as you can imagine) to assess the severity of fatigue and its impact on daily functioning. A global fatigue score is obtained by averaging all the items (1-3: mild, 4-7: moderate, 8-10: severe)
Change in Quality of life | At baseline, 6 weeks, and 12 weeks
  Quality of life collected by the EORTC Core Quality of Life Questionnaire (EORTC-QLQ-30) - a 30 question questionnaire with lower higher scores indicating a positive situation.
Sleep quality | At baseline, 6 weeks, and 12 weeks
  Will be measured by the Pittsburg Sleep Quality Index a self reported inventory to measure sleep quality. Questions are answered on 0-3 scale with higher scores indicating greater sleep pathology.
Anxiety | At baseline, 6 weeks, and 12 weeks
  The Beck Anxiety Score is a measurement on a scale from 0 to 63 obtained by using the Beck Anxiety Inventory tool to assess symptoms of anxiety. A higher score correlates to increased anxiety whereas a lower score expresses a lower amount of anxiety.
Self-reported measures of stress | At baseline, 6 weeks, and 12 weeks
  Stress will be measured by the Perceived Stress Scale. The scale measures the degree to which one perceives situations in one's life as stressful on a Likert Scale of 0 to 4 with 0 indicating never, and 4 indicating very often. Higher scores indicate higher levels of perceived stress
Self-reported measures of depression | At baseline, 6 weeks, and 12 weeks
  Will be measured by the Centers for Epidemiology Studies Depression Scale used as a screen to identify clinically significant depression; a cutoff score of greater than 16 has been shown to correlate with clinically significant depression. In addition, a score between 8 and 15 has been used to define subsyndromal depression. The possible range of scores is zero to 60, with the higher scores indicating more symptoms, weighted by frequency of occurrence during the past week.
Measures of fitness | At baseline, 6 weeks, and 12 weeks
  Will be measured with a submaximal exercise test. A 6 minute cycling exercise test.

CONTACTS AND LOCATIONS:
Overall Officials: Ellis Levine, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States